CLINICAL TRIAL: NCT00364988
Title: Combination Therapy With Pioglitazone and Losartan Provides Additional Renoprotection in Subjects With Type 2 Diabetic Nephropathy
Brief Title: Pioglitazone and Losartan Provides Additional Renoprotection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hui Min Jin, Chief,department of Nephrology,shanghai No.3 people's hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLAN
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes; Diabetic Nephropathy
Keywords: pioglitazone; losartan; proteinuria; end stage renal disease (ESRD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Proteinuria; Kidney Failure, Chronic | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pioglitazone+losartan — Pioglitazone (30 mg/daily) losartan (100 mg daily)
Drug: losartan — losartan (100 mg daily)

SUMMARY:
Peroxisomal proliferator-activated receptor agonist pioglitazone and rosiglitazone are currently used in the treatment of type 2 diabetes, as efficient insulin sensitizers alone or in combination with insulin.angiotensin II receptor antagonist losartan reduced the levels of proteinuria.Whether Combination therapy with pioglitazone and losartan provides additional renoprotection in subjects with type 2 diabetic nephropathy,it's worth researching.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose (FPG) level of 3.3-9.0mmol/L
* 2h plasma glucose level of 7.5-13 mmol/L
* serum creatinine values between 190 and 660umol/L
* Two occasions of a ratio of urinary albumin to urinary creatinine≥300 or 24 hours urinary protein concentration is >150mg
* Informed consent

Exclusion Criteria:

* Type1 diabetes or nondiabetic renal disease
* abnormal liver function
* heart dysfunction

Ages: 32 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Renal function | 12 month
  fasting glucose, HbA 1c , Scr, 24-hour urinary protein excretion, and endogenous creatinine clearance (Ccr)

CONTACTS AND LOCATIONS:
Overall Officials: Hui M Jin, MD, Principal Investigator — Shanghai No.3 People's Hospital